CLINICAL TRIAL: NCT02481089
Title: Polymorphisms in Key Genes of Glycolytic Pathway: Influence on Radiosensitivity in Nasopharyngeal Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hunan Province Tumor Hospital (Other)
Responsible Party: Principal Investigator, Hui Wang, chief of thoracic radiation oncology department, Hunan Province Tumor Hospital
Other Study IDs: warburg snp
Record Dates: First submitted 2015-06-02; First posted 2015-06-25 (Estimated); Last update posted 2016-02-19 (Estimated); Status verified 2016-02

CONDITIONS: Nasopharyngeal Carcinoma; Single Nucleotide Polymorphisms; Radiosensitivity
MeSH Terms: conditions — Nasopharyngeal Carcinoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- training group
  Interventions: Other: validation group

INTERVENTIONS:
Other: validation group

SUMMARY:
Warburg effect is an important feature of tumors,and genetic variation is one of the main factors of individual differences to radiotherapy treatment response for nasopharyngeal carcinoma(NPC). Through the previous work investigators found that the p53 codon72 (Pro/Arg) was related to the prognosis of NPC; Using the method of proteomics, investigators discovered glycolysis related gene such as PGK1, ALDOA，was associated with radiosensitivity.Thus,with all the previous work,investigators hypothesize that the key gene polymorphisms in glycolytic pathway, such as p53 , influence the glycolytic pathway,which leads to differences in radiosensitivity of NPC. This projects will include 600 cases of patients with NPC to detect common glycolytic key genes polymorphisms. Besides,investigators correlate these factors with their radiosensitivity and prognosis.Then, prediction model will be established, and validation of the prediction model will be done. Using enzyme-labeling instrument ，comet assay and clonogenic assay，cytological experiments will further investigate the influence of key gene polymorphisms on the glycolysis efficiency and mechanism of radiation sensitivity.Thus,investigators could provide theoretical basis of individualized treatment for NPC.

ELIGIBILITY:
Inclusion Criteria:

* pathological identified NPC
* KPS≥70
* tolerable and agree for IMRT and concurrent chemotherapy
* without severe other diseases
* informed consent

Exclusion Criteria:

* reject treatment
* cannot tolerate the treatment
* distant metastasis before treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: npc patients who can tolerable and agree for IMRT and concurrent chemotherapy
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2015-06; Primary Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
progression free survival | up to 60 months

CONTACTS AND LOCATIONS:
Locations (1):
- Hunan province tumor pospital, Changsha, Hunan, China